CLINICAL TRIAL: NCT00002378
Title: A Randomized Phase IIIB Comparative Study to Evaluate Saquinavir Soft Gel Capsule (SGC) TID Regimen in Combination With Two NRTIs Versus Saquinavir Soft Gel Capsule (SGC) BID Regimen in Combination With Two NRTIs Versus Saquinavir Soft Gel Capsule (SGC) BID Plus Nelfinavir BID Plus a NRTI in HIV-1 Infected Patients
Brief Title: A Comparison of Three Anti-HIV Drug Combinations Containing Saquinavir Soft Gelatin Capsules Used in HIV-1 Infected Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 229H; NR15520; M6101
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1998-12

CONDITIONS: HIV Infections
Keywords: HIV-1; Drug Therapy, Combination; Zidovudine; Stavudine; HIV Protease Inhibitors; Lamivudine; RNA, Viral; Dosage Forms; Saquinavir; Reverse Transcriptase Inhibitors; Anti-HIV Agents; Viral Load; Nelfinavir
MeSH Terms: conditions — HIV Infections | interventions — Ritonavir; Nelfinavir; Saquinavir; Delavirdine; Lamivudine; Stavudine; Zidovudine

INTERVENTIONS:
Drug: Ritonavir
Drug: Nelfinavir mesylate
Drug: Saquinavir
Drug: Delavirdine mesylate
Drug: Lamivudine
Drug: Stavudine
Drug: Zidovudine

SUMMARY:
To determine the proportion of patients whose plasma HIV-1 RNA level falls below the level of detection (< 400 copies/ml) at week 24 of study therapy. To determine the absolute change in plasma HIV-1 RNA during the 24 weeks of study treatment. To collect safety data on the treatment regimens.

AS PER AMENDMENT 12/12/97: To compare the virologic response of Fortovase (FTV) (Saquinavir) Soft Gel Capsule (SGC) tid plus nucleoside reverse transcriptase inhibitors (NRTIs) versus FTV bid plus NRTIs. Further, to compare the virologic response of FTV tid plus NRTIs versus FTV bid plus Nelfinavir bid plus a NRTI with respect to: the percentage of patients whose plasma HIV-1 RNA level falls below the Amplicor assay level of detection (< 400 copies/ml) at week 24 and week 48.

DETAILED DESCRIPTION:
Patients will be randomized to receive 1 of 3 study regimens: Group A - Saquinavir (SQV) sgc plus 2 new reverse transcriptase inhibitors (RTIs), Group B - SQV sgc plus delavirdine plus new RTI, and Group C - SQV sgc plus nelfinavir plus new RTI, or SQV sgc plus ritonavir plus 2 new RTIs.

NOTE: "New RTI" is defined for this study as any reverse transcriptase inhibitor to which the patient has never been exposed.

AS PER AMENDMENT 12/12/97: In this open-label, multicenter, Phase IIIB, comparative study, 825 patients are randomized to treatment arms. (NOTE: 50% of the patients will be treatment naive and 50% will be NRTI experienced.) Further, patients are randomized with stratification based on HIV-1 RNA level (5,000-30,000 copies/ml vs. greater than 30,000 copies/ml) and prior antiretroviral therapy to one of the three study arms.

The drug regimens for the three treatment arms are as follows:

ARM A: Fortovase (FTV), plus 2 new NRTIs*. ARM B: FTV plus 2 new NRTIs*. ARM C: FTV plus nelfinavir plus new NRTI**.

* Naive patients in Arm A and Arm B will take: d4T (or zidovudine) plus 3TC unless contraindicated.

  ** Naive patients in Arm C will take: d4T, unless contraindicated.
* NRTI experienced patients in Arms A & B should be treated with 2 NRTIs to which he/she has not been previously exposed. If the patient has only 1 NRTI to which he/she has never been exposed, then the second NRTI can be one that the patient has been previously exposed to from the most distant past.

Therapy is administered for an initial 24 weeks and may be extended for an additional 24 weeks.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* HIV-1 infection.
* HIV RNA >= 5000 copies/ml by Amplicor assay.
* Signed, informed consent from parent or legal guardian for patients less than 18 years old.

Prior Medication:

Required:

(Note:

* 50% of the patients will be treatment naive).
* > 3 months cumulative therapy with antiretrovirals other than non-nucleoside reverse transcriptase inhibitors and/or protease inhibitors.
* Stable antiretroviral therapy for at least 4 weeks prior to enrollment.

Allowed:

* <= 2 weeks cumulative treatment with protease inhibitors.

AS PER AMENDMENT 12/12/97:

Required:

NRTI experienced patients:

* > 3 months cumulative therapy with antiretrovirals.
* <= 2 weeks cumulative previous treatment with non-nucleoside analogue reverse transcriptase inhibitors (NNRTIs).
* <= 2 weeks cumulative previous treatment with protease inhibitors.
* Must have at least one NRTI (preferably two) to which he/she has not been previously exposed.
* Stable antiretroviral therapy defined as within (+/-) 1 log HIV-1 RNA between the 2 most recent values greater than 8 weeks apart (may include screening visit) prior to study enrollment. (NOTE:
* If patient does not have a previous HIV-1 RNA value, screening will be accepted.)

Required:

* Note:
* 50% of the patients will be treatment naive and 50% will be NRTI experienced. AS PER AMENDMENT 12/12/97.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 825

CONTACTS AND LOCATIONS:
Locations (101):
- United States (96):
  - ASC Inc, Anniston, Alabama
  - CIGNA, Phoenix, Arizona
  - Arizona Clinical Research Ctr Inc, Tucson, Arizona
  - Univ of Arizona, Tucson, Arizona
  - Alta Bates Med Ctr, Berkeley, California
  - Ctr for Special Immunology, Irvington District, California
  - AIDS Healthcare Foundation Labs, Los Angeles, California
  - Beer Med Group, Los Angeles, California
  - Dr Charles Farthing, Los Angeles, California
  - Gottlieb Med Group, North Hollywood, California
  - Dr Wilbert Jordan, Paramount, California
  - AIDS Community Research Consortium, Redwood City, California
  - Dr Daniel Pearce, San Francisco, California
  - UCSF - San Francisco Gen Hosp, San Francisco, California
  - Kaiser Permanente Med Ctr, San Francisco, California
  - QUEST Clinical Research, San Francisco, California
  - Marin County Specialty Clinic, San Rafael, California
  - Shared Med Research Foundation, Tarzana, California
  - Denver Public Health Dept / Disease Control Services, Denver, Colorado
  - Kaiser Permanente, Infectious Disease, Denver, Colorado
  - Georgetown Univ Med Ctr, Washington D.C., District of Columbia
  - Anderson Clinical Research, Washington D.C., District of Columbia
  - Providence Hosp, Washington D.C., District of Columbia
  - IDC Research Initiative, Altamonte Springs, Florida
  - Urgent Care Ctr, Fort Lauderdale, Florida
  - Stratogen of Ft Lauderdale, Fort Lauderdale, Florida
  - Dr Robert Schwartz, Fort Myers, Florida
  - Duval County Health Dept, Jacksonville, Florida
  - Steinhart Medical Associates, Miami, Florida
  - Stratogen Health of Palm Beach, Palm Beach Gardens, Florida
  - Ctr for Quality Care, Tampa, Florida
  - Univ of South Florida, Tampa, Florida
  - Infectious Disease Research Institute Inc, Tampa, Florida
  - Treasure Coast Infectious Disease Consultants, Vero Beach, Florida
  - AIDS Research Consortium of Atlanta, Atlanta, Georgia
  - Infectious Disease Specialists of Atlanta, Decatur, Georgia
  - Northwestern Univ Med Ctr, Chicago, Illinois
  - SIU School of Medicine, Springfield, Illinois
  - Carle Clinic Association, Urbana, Illinois
  - Indiana Univ Hosp, Indianapolis, Indiana
  - Univ of Kentucky / Kentucky Clinic Annex #, Lexington, Kentucky
  - Community Research Initiative, Brookline, Massachusetts
  - Univ of Massachusetts Med Ctr, Worcester, Massachusetts
  - Harper Hosp, Detroit, Michigan
  - Saint Joseph's / Mercy Hosp, Ypsilanti, Michigan
  - Abbott Northwestern Hosp, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Univ of Missouri at Kansas City School of Medicine, Kansas City, Missouri
  - Antibiotic Research Associates, Kansas City, Missouri
  - HIV Wellness Ctr / Univ Med Ctr, Las Vegas, Nevada
  - Dartmouth-Hitchcock Med Ctr, Lebanon, New Hampshire
  - UMDNJ - New Jersey Med School / Cooper Hosp, Camden, New Jersey
  - VAMC New Jersey Healthcare System, East Orange, New Jersey
  - New Jersey Community Research Initiative, Newark, New Jersey
  - St Joseph's Hosp & Med Center, Paterson, New Jersey
  - Albany Med College / Division of HIV Medicine A158, Albany, New York
  - Brookdale Univ Med Ctr, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Nassau County Med Ctr, East Meadow, New York
  - Elmhurst Hosp, Elmhurst, New York
  - North Shore Univ Hosp, Manhasset, New York
  - Mt Vernon Hosp, Mount Vernon, New York
  - Dr Michael Mullen, New York, New York
  - Peter Krueger Clinic, New York, New York
  - Howard Grossman, New York, New York
  - AIDS Clinical Trials Unit, New York, New York
  - Dr Douglas Dieterich, New York, New York
  - Dr Ron Grossman, New York, New York
  - Liberty Med Group, New York, New York
  - St Lukes / Roosevelt Hosp / HIV Center, New York, New York
  - New York / Cornell Med Ctr, New York, New York
  - New York Hosp - Cornell Med Ctr, New York, New York
  - New York Hosp / Cornell Med Ctr, New York, New York
  - Harlem Hosp Ctr, New York, New York
  - Montefiore Med Ctr, The Bronx, New York
  - Carolinas Research Associates, Charlotte, North Carolina
  - Nalle Clinic, Charlotte, North Carolina
  - East Carolina Univ School of Medicine, Greenville, North Carolina
  - Bowman Gray School of Medicine, Winston-Salem, North Carolina
  - Univ of Cincinnati Med Ctr / Holmes Division, Cincinnati, Ohio
  - Oklahoma Univ Health Science Ctr, Oklahoma City, Oklahoma
  - Lehigh Valley Hosp, Allentown, Pennsylvania
  - Allegheny Univ Hosp, Philadelphia, Pennsylvania
  - Dr Jay Kostman, Philadelphia, Pennsylvania
  - Roger Williams Med Ctr, Providence, Rhode Island
  - Burnside Clinic, Columbia, South Carolina
  - Austin Infectious Disease Consultants, Austin, Texas
  - Dr Nicholaos Bellos, Dallas, Texas
  - Univ of Texas Southwestern Med Ctr of Dallas, Dallas, Texas
  - North Texas Infectious Disease Consultants, Dallas, Texas
  - Houston Clinical Research Network, Houston, Texas
  - ONCOL Med Associates / PA, Houston, Texas
  - Houston Med Ctr, Houston, Texas
  - Infectious Disease Physicians Inc, Annandale, Virginia
  - Swedish Med Ctr / Dr Peter Shalit, Seattle, Washington
  - Aurora Med Group, Milwaukee, Wisconsin
- Medizinische Einrichtungen der Heinrich U, Düsseldorf, Germany
- Ospedale S Raffaele, Milan, Italy
- San Juan Veterans Administration Med Ctr, San Juan, Puerto Rico
- Hosp Valle D Hebron, Barcelona, Spain
- Royal Liverpool Univ Hosp, Liverpool, United Kingdom